CLINICAL TRIAL: NCT00252590
Title: Health Focused Motivational Treatment for Alcohol Dependent Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEUA-003-05S
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Alcoholism
Keywords: Psychotherapy motivational intervention
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Health Motivational Feedback (Experimental): Personalized health-related feedback
  Interventions: Behavioral: Health Motivational Feedback
- Health Education (Active Comparator): Non-personalized didactic health-related education
  Interventions: Behavioral: Health Education
- Control - treatment as usual (Active Comparator): No added treatment control
  Interventions: Behavioral: Control - treatment as usual

INTERVENTIONS:
Behavioral: Health Motivational Feedback — Personalized feedback on health status
  Arms: Health Motivational Feedback
Behavioral: Health Education — Generalized health education related to alcohol use
  Arms: Health Education
Behavioral: Control - treatment as usual — Control group with no additional intervention
  Arms: Control - treatment as usual

SUMMARY:
The purpose of this study is to determine whether a health focused motivational intervention will reduce alcohol use for dependent veterans who are receiving outpatient alcohol and drug treatment.

DETAILED DESCRIPTION:
The early months of addiction treatment are a high risk time for relapse. The purpose of this study is to examine whether a health-related intervention delivered in an individual session with a therapist once per month in the initial 4 months of addiction treatment will reduce alcohol use among veterans already enrolled in weekly outpatient treatment group at the VA San Diego Healthcare System. In order to answer this question, study participants will be randomly assigned to one of three study conditions: 1) The Health Motivational condition that receives individual personalized health feedback and motivational activities, 2) the Health Education condition that receives individual education about health problems associated with the heavy alcohol use, and 3) the treatment as usual group that will receive no additional treatment. All participants will be assessed on a monthly basis for 4 months to evaluate alcohol use, drug use, and health status.

ELIGIBILITY:
Inclusion Criteria:

- Veterans receiving outpatient treatment at the VA San Diego Healthcare System Alcohol and Drug Treatment Program for a diagnosis of Alcohol Dependence

Exclusion Criteria:

* Diagnosis of Bipolar Disorder or Psychotic Disorder.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2005-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Tate, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego
Locations (1):
- VA San Diego Healthcare System, San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Motivational Feedback: Personalized health-related feedback
  Health Motivational Feedback: Personalized feedback on health status provided in four once monthly 45 minute sessions. Information for feedback was attained with assessments and blood serum testing.
- Health Education: Non-personalized didactic health-related education
  Health Education: Generalized health education related to alcohol use provided in four once monthly 45-minute sessions. Topics for sessions include sleep, pain, cardiovascular health, and gastrointestinal health.
Period: Overall Study
Arm/Group | Health Motivational Feedback | Health Education | Control - Treatment as Usual
Started | 35 | 30 | 34
Completed | 33 | 28 | 31
Not Completed | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Motivational Feedback | Health Education | Control - Treatment as Usual | Total
Number analyzed (Participants) | 35 | 30 | 34 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (11.0) | 49.4 (8.2) | 49.1 (11.7) | 48.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 9
  Male | 31 | 27 | 32 | 90
Region of Enrollment [Number; unit: participants]
  United States | 35 | 30 | 34 | 99
Percentage Days Abstinent all substances [Mean (Standard Deviation); unit: percentage] | 48.6 (31.5) | 59.6 (32.0) | 47.4 (29.2) | 51.5 (31.0)
Percentage Days Abstinent alcohol [Mean (Standard Deviation); unit: percentage] | 49.1 (31.0) | 60.1 (31.9) | 48.2 (28.8) | 52.1 (30.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days Abstinent From Alcohol
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of days abstinent alcohol
Arm/Group | Health Motivational Feedback | Health Education | Control - Treatment as Usual
Number analyzed (Participants) | 33 | 28 | 31
percentage of days abstinent alcohol | 91.4 (14.2) | 87.3 (23.6) | 83.0 (26.8)
Statistical Analysis 1: Comparison: Health Motivational Feedback vs Health Education vs Control - Treatment as Usual; Test type: Superiority or Other; p = 0.32, ANOVA

2. Secondary Outcome: Percentage of Days Abstinent From All Substances
Description: Percentage of days abstinent from both alcohol and drugs
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of days abstinent
Arm/Group | Health Motivational Feedback | Health Education | Control - Treatment as Usual
Number analyzed (Participants) | 33 | 28 | 31
percentage of days abstinent | 91.2 (14.2) | 84.1 (27.8) | 82.1 (26.7)

ADVERSE EVENTS:
Time Frame: 3 years, 8 months
Arm/Group | Health Motivational Feedback | Health Education | Control - Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/30 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/30 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Motivational Feedback (N=35) | Health Education (N=30) | Control - Treatment as Usual (N=34)
Inpatient psychiatric hospital admission (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Treatment for increased psychiatric symptoms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No